CLINICAL TRIAL: NCT01072162
Title: A Randomized, Open-label, Five-period, Balanced Crossover Study to Evaluate the Relative Bioavailability of an Eltrombopag Powder for Oral Suspension (PfOS) Formulation Relative to the Commercial 25 mg Tablet Formulation and to Evaluate Administration of the PfOS Formulation With and Separated 2 Hours From a High Calcium Meal in Healthy Adult Subjects
Brief Title: Relative Bioavailibilty for Pediatric Powder for Suspension (PfOS) Formulation and Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 111718
Record Dates: First submitted 2010-02-12; First posted 2010-02-19 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: healthy; powder for suspension; tablets; bioavailibility; eltrombopag
MeSH Terms: conditions — Purpura | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm B (Experimental): 25 mg powder for oral suspension single dose fasted.
  Interventions: Drug: Eltrombopag
- Arm C (Experimental): 25 mg powder for oral suspension administered with a meal
  Interventions: Drug: Eltrombopag
- Arm D (Experimental): 25 mg powder for oral suspension administered 2 hours prior to meal
  Interventions: Drug: Eltrombopag
- Arm E (Experimental): 25 mg powder for oral suspension administered 2 hours after to meal
  Interventions: Drug: Eltrombopag
- Arm A (Other): Commercially available eltrombopag 25 mg tablet
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — 25 mg tablet
  Arms: Arm A
Drug: Eltrombopag — 25 mg powder for oral suspension
  Arms: Arm B; Arm C; Arm D; Arm E

SUMMARY:
This is a randomized, open-label, five-period, balanced crossover study conducted in approximately 40 healthy adult subjects enrolled at one study center in the USA. Subjects receive five eltrombopag treatments: tablet fasted, Powder for Oral Suspension (PfOS) fasted, PfOS with a high calcium meal, PfOS 2 hours prior to a high calcium meal, and PfOS 2 hours after a high calcium meal, and each treatment is a single 25 mg dose. There is a 10 to 14 day washout between periods, and between the last dose of study drug and the follow-up visit. During each treatment period, subjects undergo serial PK sampling over 72 hours for measurement of plasma eltrombopag concentrations. Safety is assessed by vital signs, clinical safety laboratory assessments, and adverse events reporting.

DETAILED DESCRIPTION:
This is a randomized, open-label, five-period, balanced crossover study conducted in approximately 40 healthy adult subjects enrolled at one study center in the USA. Subjects receive five eltrombopag treatments: tablet fasted, PfOS fasted, PfOS with a high calcium meal, PfOS 2 hours prior to a high calcium meal, and PfOS 2 hours after a high calcium meal, and each treatment is a single 25 mg dose. There is a 10 to 14 day washout between periods, and between the last dose of study drug and the follow-up visit. During each treatment period, subjects undergo serial PK sampling over 72 hours for measurement of plasma eltrombopag concentrations. Safety is assessed by vital signs, clinical safety laboratory assessments, and adverse events reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects with no clinically significant abnormality identified by physician by evaluation of medical history, physical examination, clinical laboratory tests or electrocardiogram (ECG).
2. Male and female subjects between the ages of 18 to 64 years of age inclusive, at the time of signing the informed consent.
3. Subject is able to understand and comply with the protocol requirements, instructions and restrictions.
4. Capable of giving written informed consent which includes compliance with the requirements and restrictions listed in the consent form.
5. Body weight ≥ 50kg (110 lbs) for men and ≥ 45 kg (99 lbs) for women and body mass index (BMI) of 18.5 to 29.9 kg/m2 inclusive.
6. A platelet count within normal range and not > 400,000 plt/uL.
7. Male subjects, who are not surgically sterile, must agree on abstinence or to use a double barrier method, such as, a condom plus spermicidal agent (foam/gel/film/cream/suppository). This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of medication.
8. A female subject is eligible to participate if she is neither pregnant nor lactating, and falls into one of the following categories:

   * non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or bilateral oophorectomy, or post-menopausal females defined as being amenorrheic for greater than one year and having serum estradiol and follicle stimulating hormone levels consistent with menopause.
   * child-bearing potential with negative beta human chorionic gonadotropin (beta/hCG) test and agrees to comply with recognized non-hormonal contraceptive methods from screening or at least two weeks prior to first dose (whichever is earlier) until the follow-up visit. Recognized non-hormonal contraceptive methods include: complete abstinence from intercourse, male partner sterilization, two forms of barrier contraception (e.g. condom and occlusive cap (diaphragm or cervical/vault caps with spermicide), or intrauterine device (IUD), or intrauterine system (IUS) with a < 1% failure rate stated in the product label.

Exclusion Criteria:

1. History of Gilbert's syndrome.
2. Any previous history of deep vein thrombosis or any other thromboembolic event.
3. History of thrombocytopenia or bleeding due to abnormal platelet number or function.
4. Clotting factor abnormalities associated with hypercoagulability, specifically Factor V Leiden, Protein C or Protein S deficiency or antithrombin III deficiency.
5. Elevated blood pressure (BP) at screening (systolic > 140 mm Hg, diastolic > 85 mm Hg). If the subject's BP is elevated on the first measurement, complete two additional BP measurements two minutes apart and average the three assessments to evaluate this criteria. If averaged BP exceeds the safety criteria, the subject should be excluded.
6. History of atrial fibrillation, mitral valve prolapse, significant heart murmur or vascular bruit.
7. Prolonged QTc interval (Bazett's) at screening (for females > 450 msec and for males > 430 msec). If the QTc interval is prolonged on the initial ECG, then complete two additional ECGs 5 minutes apart and take the average QTc measurements of all three ECGs to evaluate this criteria. If averaged QTc exceeds the safety criteria, the subject should be excluded.
8. Female subjects currently receiving hormone replacement therapy (HRT).
9. Positive for HIV, hepatitis B virus or hepatitis C virus assays at screening.
10. Positive urine drug screen including alcohol at screening or pre-dose (Day -1).
11. History of alcohol/drug abuse or dependence within 12 months of the study.
12. History of alcohol consumption in the past six months exceeding 7 units/week for women and 14 units/week for men (where 1 unit = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor).
13. Urinary cotinine levels indicative of smoking at screening or pre-dose (Day -1). History of regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
14. Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
15. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
16. Use of prescription or non-prescription drugs (including aspirin and non-steroidal anti-inflammatory drugs [NSAIDs]), vitamins, herbal and dietary supplements within seven days (or 14 days if the drug is a potential enzyme inducer, such as St. John's Wort) or five half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
17. Subjects who have donated plasma within seven days prior to the screening visit or where participation in this study would result in donation of blood in excess of 500 mL within a 56-day period.
18. History of sensitivity to any of the study medications, or components thereof.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01-12 (Actual); Primary Completion 2010-04-07 (Actual); Study Completion 2010-04-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the relative bioavailability of a PfOS formulation relative to the commercial eltrombopag 25 mg tablet formulation in healthy adult subjects. | 72 hours x 2 periods
Evaluate the effect of a high calcium, moderate fat and calorie meal on the pharmacokinetics of a single oral 25 mg dose of eltrombopag PfOS in healthy adult subjects when eltrombopag is administered concurrently, two hours before, or two hours afte | 72 hours x 3 periods

SECONDARY OUTCOMES:
Assess the safety and tolerability of single oral doses of eltrombopag. | 12-14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Background] Wire MB, Bruce J, Gauvin J, Pendry CJ, McGuire S, Qian Y, Brainsky A. A randomized, open-label, 5-period, balanced crossover study to evaluate the relative bioavailability of eltrombopag powder for oral suspension (PfOS) and tablet formulations and the effect of a high-calcium meal on eltrombopag pharmacokinetics when administered with or 2 hours before or after PfOS. Clin Ther. 2012 Mar;34(3):699-709. doi: 10.1016/j.clinthera.2012.01.011. Epub 2012 Feb 14. PMID 22336488
- See also: Results for study 111718 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111718?search=study&study_ids=111718#rs